CLINICAL TRIAL: NCT00954278
Title: A Phase I, Intrapatient Dose-Escalation Study of Sorafenib in Advanced or Relapsed Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Intra-patient Dose Escalation Study of Sorafenib in Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO08511; H-2009-0011 (Other: Institutional Review Board); IST 000381; A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison); NCI-2011-00813 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2009-07-30; First posted 2009-08-07 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: non small cell lung cancer; phase 1; sorafenib; intrapatient dose escalation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib (Experimental)
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — sorafenib (400mg or 600mg or 800mg) by mouth twice daily, for 28 days
  Other Names: BAY-439006; Nexavar

SUMMARY:
The purpose of this study is to determine the number of patients with advanced, relapsed non-small cell lung cancer who can tolerate dose escalation sorafenib from 400 mg twice daily to either 600 mg twice daily or 800 mg twice daily. Safety and tolerability of sorafenib will also be examined.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is the leading cause of cancer-related mortality in the U.S. Time to progression in advanced disease remains poor and further study of newer agents with novel mechanisms of action is needed to improve duration and quality of life for NSCLC patients.

Sorafenib is an oral-multi-kinase inhibitor with effects on tumor proliferation and tumor angiogenesis. Sorafenib has demonstrated activity in preclinical models of NSCLC both in combination with chemotherapy and as monotherapy. A recent intra-patient dose escalation trial of sorafenib in renal cell carcinoma showed positive response rates and tolerability up to 1200mg in 91% of patients.

This study attempts a similar dose-escalation of sorafenib in NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, advanced (stage IIIB with pleural effusion, stage IV, or recurrent), kras mutation positive, non-small cell lung cancer (NSCLC)
* Measurable disease per RECIST criteria
* Patients must have received one + prior chemotherapy regimens for NSCLC
* Patients may have treated and clinically stable brain metastases
* Adequate bone marrow, liver and renal function
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation, and for 3 months after last administration of sorafenib
* Patients must have the ability to understand and willingness to sign a written informed consent
* International normalized ratio(INR) < 1.5 or prothrombin time/ partial thromboplastin time (PT/PTT) within normal limits

Exclusion Criteria:

* Prior exposure to a Ras pathway inhibitor
* Any other anti-tumor therapy within 3 weeks of enrollment
* Prior bevacizumab within the past 6 weeks
* An active secondary malignancy except non-melanoma skin cancer
* Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina or new onset angina or myocardial infarction within the past 6 months
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Uncontrolled hypertension, defined as systolic blood pressure > 150mm Hg or diastolic pressure > 90mm Hg, despite optical medical management
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C
* Active clinically serious infection > Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
* Thrombolic or embolic events such as cerebrovascular accident including transient ischemic attack within the past 6 months
* Pulmonary hemorrhage/bleeding event >/= CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event >/= CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug
* Use of St. John's Wort or rifampin
* Known or suspected allergy to sorafenib or any agent given in the course of the trial
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07-28 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2015-12-23 (Actual)

PRIMARY OUTCOMES:
Toleration of dose escalation (dose-limiting toxicities) | One year

SECONDARY OUTCOMES:
Safety of sorafenib in dose-escalation (adverse events and serious adverse events) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Traynor, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/